CLINICAL TRIAL: NCT00638209
Title: Insulin Sensitivity of the Brain in Pathogenesis of Diabetes Mellitus Typ 2
Brief Title: Insulin Sensitivity of the Brain in Pathogenesis of Diabetes Mellitus Type 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Prof. Andreas Fritsche, University Hospital Tuebingen, Internal Medicine IV
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MEG-KFO-2; EudraCT 2006-004734-32; KFO-114
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2008-03-19 (Estimated); Status verified 2008-03

CONDITIONS: Human Physiology of Energy Homeostasis
MeSH Terms: interventions — Insulin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Active Comparator)
  Interventions: Drug: Human insulin
- P (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Human insulin
  Arms: I
Drug: Saline
  Arms: P

SUMMARY:
The purpose of the study is to investigate whether insulin sensitivity of the human brain correlates with insulin sensitivity of the liver.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 Risk factor(s) for type 2 diabetes (e.g. overweight, family history of diabetes)

Exclusion Criteria:

* Type 2 diabetes pregnancy acute or chronic diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Insulin effect on cortical function (spectral analysis) | 2 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Tuebingen, Internal Medicine IV, Tübingen
  - University Hospital Tuebingen, Tübingen